CLINICAL TRIAL: NCT00252902
Title: Emergency Department Initiated Tobacco Treatment (EDITT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: The Cooper Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DA-16698-01; DA-16698-01
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2013-10

CONDITIONS: Tobacco Use
Keywords: tobacco; emergency department; motivation; counseling
MeSH Terms: conditions — Tobacco Use; Emergencies | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior change counseling

SUMMARY:
The primary purpose of the study is to refine the intervention protocols for two ED-initiated tobacco interventions and to assess the magnitude of the effect size that can be expected. We expect the intervention groups to have greater sustained abstinence, point-prevalence abstinence, and motivation to change when compared to the treatment as usual group at 1- and 3-month follow-up.

DETAILED DESCRIPTION:
Most surveys of emergency physicians indicate that smoking cessation counseling rarely occurs in routine clinical practice. Prochazka and colleagues (1996) studied 196 members of the Colorado Chapter of the American College of Emergency Physicians and found that only 27% reported routinely asking patients to quit smoking. We conducted a similar survey study and found that only 19% of emergency physicians practicing in an urban teaching hospital reported that they routinely counseled their tobacco using patients to quit. A study of 63 adult smokers presenting to the ED with symptoms of acute respiratory illness found that only 9% were offered any assistance with quitting (Bock et al., 2001). Clearly, more research was needed to investigate smoking interventions initiated in the ED.

Currently, not much is known about how best to intervene with smokers in the ED. This proposal describes a pilot study designed to explore two interventions. Research that expands our knowledge of ED-initiated tobacco interventions has tremendous public health potential, especially for the under-served populations that are over-represented in the ED patient population.This study is designed primarily to yield effects size parameters so a larger RCT can be planned. For this reason, it is not powered specifically to detect a given difference, but, rather, simply to provide an idea of the size of the effect so we can determine how many subjects would be needed in a future trial in order to demonstrate statistical significance and clinical utility. It will also be used to refine the study design, protocols, and treatment manuals for the future trial.

This study will be a randomized, single-blind, controlled trial that will compared two types of ED-initiated tobacco treatment to treatment-as-usual. 75 ED patients who meet all inclusion and exclusion criteria will be randomly assigned to one of three groups using a 2:2:1 ratio: Group One: Enhanced Care (n=30), Group Two: Dynamic Referral (n=30), or Group Three: Clinic Referral (n=15). This assignment ratio is being used to maximize experience with the treatments. The two interventions will be delivered by trained counselors and are described below. Baseline measures of smoking and other related variables will be taken during the ED visit. An interviewer blind to study group assignment will conduct follow-up assessments via telephone at 1- and 3-months after the ED visit. We expect a 25% attrition, yielding follow-up data at 3-months on 23, 23, and 11 patients, respectively, for each Group.

Primary outcomes will include: sustained abstinence from the ED visit to the follow-up time periods and 7-day point prevalence abstinence. Secondary outcomes will be: presence of a quit attempt >= 24 hours and readiness to change.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* receiving treatment in the ED
* smoking at least 10 cigarettes daily

Exclusion Criteria:

* too ill to participate
* temporary shelter
* no phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Sustained abstinence (from tobacco)
7-day Point prevalence abstinence
Any quit attempt >= 24 hours

SECONDARY OUTCOMES:
Motivation to quit
Treatment engagement

CONTACTS AND LOCATIONS:
Overall Officials: Edwin D Boudreaux, PhD, Principal Investigator — Cooper University Hospital, UMDNJ-Robert Wood Johnson Medical School
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

REFERENCES:
- [Result] Boudreaux ED, Baumann BM, Perry J, Marks D, Francies S, Camargo CA Jr, Ziedonis D. Emergency department initiated treatments for tobacco (EDITT): a pilot study. Ann Behav Med. 2008 Dec;36(3):314-25. doi: 10.1007/s12160-008-9066-3. Epub 2008 Dec 3. PMID 19050988